CLINICAL TRIAL: NCT07133568
Title: Design, Development, and Validation of a Recreational Exercise Intervention in Older Adults to Improve Intrinsic Capacity and Motivation: A Randomized Clinical Trial
Brief Title: Fun Exercise Intervention for Older Adults to Improve Intrinsic Capacity and Motivation
Acronym: FEXO-COM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Professor, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-77
Record Dates: First submitted 2025-07-25; First posted 2025-08-21 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-08

CONDITIONS: Sarcopenia; Frailty Syndrome
Keywords: intrinsic capacity; fun exercise; playful exercise; frailty; multicomponent exercise; otago
MeSH Terms: conditions — Sarcopenia; Frailty | interventions — Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FEXO (Fun EXercise for Older adults) (Experimental): Participants assigned to the experimental group will take part in a structured multicomponent exercise program specifically designed for older adults. The program, named FEXO, emphasizes recreational and motivational aspects to enhance adherence and enjoyment. It consists of three non-consecutive 1-hour sessions per week for 14 weeks. Exercises are conducted in a group setting (maximum ratio 1 instructor to 15 participants) and are progressively adapted according to the functional capacity of each participant, assessed using the Short Physical Performance Battery (SPPB).
  The program uses simple, low-cost, portable materials such as elastic bands, chairs, soft balls, scarves, maracas, and a bubble machine, creating a playful and inclusive environment.
  Interventions: Other: Fun Exercise for Older Adults (FEXO)
- OTAGO multicomponent exercise program (Active Comparator): Participants in the control group will follow the OTAGO Exercise Program, a widely studied and evidence-based intervention aimed at reducing fall risk and improving lower-limb strength and balance in older adults. This program also lasts 14 weeks, with three non-consecutive sessions per week, delivered in a group format under the supervision of a physiotherapist.
  Unlike the FEXO program, OTAGO is more traditional and does not include recreational or cognitive stimulation elements. It serves as an active comparator to evaluate whether incorporating fun and motivational strategies improves adherence, engagement, and intrinsic capacity.
  Interventions: Other: OTAGO

INTERVENTIONS:
Other: Fun Exercise for Older Adults (FEXO) — The FEXO (Fun Exercise for Older Adults) program is a 14-week, multicomponent, recreational exercise intervention designed to enhance intrinsic capacity, motivation, and adherence in community-dwelling older adults. Participants engage in three non-consecutive, supervised group sessions per week (maximum instructor-to-participant ratio 1:15), each lasting approximately 60 minutes. The program begins with a two-week familiarization phase followed by three progressive phases (4 weeks each), with exercise intensity, repetitions, and resistance levels adjusted based on functional performance assessed by the Short Physical Performance Battery (SPPB).
  Arms: FEXO (Fun EXercise for Older adults)
Other: OTAGO — The OTAGO Exercise Program is a structured, evidence-based intervention developed to improve lower-limb strength and balance and reduce fall risk in older adults. In this study, participants in the control group will complete three non-consecutive, supervised sessions per week for a total duration of 14 weeks. Sessions will be delivered in group settings under the supervision of a licensed physiotherapist. The program includes individualized strength training for the lower extremities, progressive balance exercises, and walking routines. Although originally designed as a home-based program, in this trial it will be implemented in indoor, climate-controlled, non-slip-floor facilities provided by local institutions. The OTAGO protocol does not include recreational, cognitive, or playful components, serving instead as a standard, structured intervention against which the FEXO program will be compared.
  Arms: OTAGO multicomponent exercise program

SUMMARY:
This randomized clinical trial aims to evaluate the effectiveness of a structured, multicomponent recreational exercise program (FEXO: Fun Exercise for Older Adults) in improving intrinsic capacity, motivation, and adherence among community-dwelling older adults. Participants aged 60 years and older will be randomly allocated to either the FEXO group or a control group performing the established OTAGO program. The intervention will last 14 weeks, with three weekly sessions. Assessments will be conducted at baseline, post-intervention, and after a 3-month follow-up.

DETAILED DESCRIPTION:
The global increase in the aging population poses significant public health and societal challenges, particularly regarding multimorbidity, frailty, and functional decline. In response, the World Health Organization has introduced the concept of Intrinsic Capacity (IC), which encompasses the physical and mental capacities an individual can draw upon. IC includes five domains: locomotion, vitality, cognition, psychological well-being, and sensory function.

Evidence supports multicomponent exercise as a primary strategy to promote healthy aging and preserve functionality in older adults. However, low adherence and motivation remain critical barriers. This study proposes a novel, recreationally oriented multicomponent program-FEXO-designed to increase engagement through fun, low-cost, group-based sessions adapted to functional levels.

The study is a two-arm, parallel-group, randomized clinical trial with a 2:1 allocation ratio (intervention:control). A total of 122 older adults from the community will be recruited and randomized into either the FEXO group or the control group (OTAGO program). Both interventions include three non-consecutive weekly sessions over 14 weeks. The FEXO program includes a familiarization phase and progressive intensity adjustments.

Sessions integrate strength, balance, coordination, cognitive stimulation, and relaxation in a recreational format using music, elastic bands, and playful materials. Primary outcomes include changes in Intrinsic Capacity, assessed through standardized tools across its five domains. Secondary outcomes include anthropometric data, cardiovascular parameters, physical performance tests, cognitive function, depression, resilience, and exercise motivation. Adherence will be tracked as the percentage of sessions attended.

Statistical analysis will be conducted on an intention-to-treat basis using two-way ANOVA, with effect sizes and confidence intervals reported. The study has been approved by the Ethics Committee of CEU Cardenal Herrera University and complies with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults aged 60 years or older.
* Able to walk independently, with or without assistive devices (e.g., cane or walker).
* Provide written informed consent before participation.
* Willing and able to attend scheduled exercise sessions and assessments over the full duration of the study.

Exclusion Criteria:

* Presence of severe psychiatric or psychological disorders that may interfere with participation or adherence.
* Physical incapacity to perform moderate-intensity exercise safely.
* Participation in another structured multicomponent exercise program during the intervention period.
* Cognitive impairment that limits comprehension or execution of instructions, as determined by clinical evaluation.
* Recent fractures, or uncontrolled cardiovascular conditions that contraindicate exercise.
* Any medical condition judged by the investigators to contraindicate physical exercise or to pose an unacceptable risk.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Intrinsic Capacity | Before and inmediately after the intervention
  It is a multidimensional concept defined by the World Health Organization to represent the total physical and mental capacities of an individual. It includes five domains: locomotion (SPPB), vitality (MDA), cognition (MMSE), psychological well-being (CSDD), and sensory function (Self-reported). Each domain contributes up to 2 points, for a total composite score ranging from 0 to 10. Higher scores indicate better intrinsic capacity and functional reserve. The specific instruments used to assess each domain are standard, validated tools, and although they contribute to the IC score, they will also be analyzed separately as secondary outcomes to better understand changes in each specific domain.
Adherence to intervention | During intervention
  Adherence will be calculated as the percentage of sessions attended out of the total planned (42 sessions over 14 weeks). Higher adherence rates reflect better feasibility and acceptance of the exercise program.
Motivation (Behavioral Regulation in Exercise Questionnaire (BREQ-3)) | Before and inmediately after the intervention
  This self-report questionnaire assesses different types of motivation toward exercise (intrinsic, identified, introjected, external, and amotivation) based on Self-Determination Theory. Each subscale ranges from 0 to 12 points. Higher scores in intrinsic and identified motivation are considered positive indicators of adherence and engagement, whereas higher scores in introjected, external, and amotivation reflect lower quality motivation and are considered unfavorable.

SECONDARY OUTCOMES:
Blood pressure | Before and inmediately after the intervention
  Resting systolic and diastolic blood pressure will be measured at all three time points using an automated sphygmomanometer, following the European Society of Hypertension guidelines. A reduction or maintenance within normal ranges (<130/80 mmHg) is considered a favorable outcome, while elevated values or increases over time indicate an unfavorable outcome.
Heart rate | Before and inmediately after the intervention
  Resting heart rate (beats per minute) will be assessed at all three time points using an automated sphygmomanometer, following the European Society of Hypertension guidelines. A reduction or maintenance within normal ranges (60-80 bpm) is considered a favorable outcome, whereas elevated resting heart rate (>80 bpm) or increases across assessments are considered unfavorable.
Frailty status (Fried criteria) | Before and inmediately after the intervention
  Frailty status will be assessed using Fried's phenotype, which classifies participants as robust (0 criteria), pre-frail (1-2 criteria), or frail (3-5 criteria) based on five components: unintentional weight loss, exhaustion, low physical activity, slow gait speed, and weak grip strength. Improvement is defined as transition to a lower frailty category (e.g., from frail to pre-frail).
Grip Strenght (JAMAR Dynamometer) | Before and inmediately after the intervention
  Grip strength will be measured using a JAMAR hand dynamometer, with participants seated, the elbow at 90°, forearm in a neutral position, and wrist slightly extended. The best of three trials is recorded in kilograms. Grip strength is a core indicator of sarcopenia and a strong predictor of functional decline, morbidity, and mortality. Higher values reflect better upper-limb muscle strength.
10-Meter Walk Test (10-MWT) | Before and inmediately after the intervention
  Participants will perform two walking trials over 10 meters: one at habitual pace and one at maximum pace. The time to walk the central 6-meter portion is recorded and converted into meters per second (m/s). Gait speed is a validated marker of frailty, physical function, and fall risk. Higher walking speeds reflect better functional status.
Mini-Mental State Examination (MMSE) | Before and inmediately after the intervention
  The MMSE evaluates general cognitive status through domains including orientation, memory, attention, language, and visuospatial skills. It yields a score from 0 to 30, with higher scores indicating better cognitive function. It is widely used for screening and monitoring cognitive impairment in older adults.
Mini Nutritional Assessment (MNA) | Before and inmediately after the intervention
  The MNA is a validated tool for detecting malnutrition or risk of malnutrition in older adults. It includes 18 items covering anthropometry, general health, dietary intake, and subjective assessment. Total scores range from 0 to 30: scores ≥24 indicate normal nutrition, 17-23.5 suggest risk of malnutrition, and <17 indicate malnutrition. Higher scores reflect better nutritional status.
Geriatric Depression Scale (GDS) | Before and inmediately after the intervention
  The Geriatric Depression Scale short form (15 items) will be used to screen for depressive symptoms in participants. Responses are binary (yes/no), and total scores range from 0 to 15. A score of 0 indicates no depressive symptoms (best psychological well-being), while 15 indicates the maximum level of depressive symptoms. Scores >5 may indicate clinical depression.
Berg Balance Scale (BBS) | Before and inmediately after the intervention
  This 14-item scale assesses balance and postural control in older adults. Each task (e.g., standing, reaching, turning) is scored from 0 (unable) to 4 (independent), with a total score ranging from 0 to 56. Scores below 45 suggest increased fall risk. Higher scores reflect better balance.
Sit-to-Stand Test (STS-5) | Before and inmediately after the intervention
  The Five-Times Sit-to-Stand test evaluates lower-limb strength and endurance. The time in seconds to complete five sit-to-stand repetitions without arm support is measured. Shorter times reflect better muscle function and physical performance.
Timed Up and Go (TUG) - Standard version | Before and inmediately after the intervention
  The standard Timed Up and Go (TUG) test is a widely used functional assessment that measures basic mobility and dynamic balance. Participants are instructed to stand up from a standard-height chair, walk a distance of 3 meters, turn around, return to the chair, and sit down. The total time required to complete the task is recorded in seconds. Shorter times indicate better functional mobility and lower risk of falls.
Trail Making Test - Part A | Before and inmediately after the intervention
  This test measures visual attention, processing speed, and cognitive flexibility. Participants are instructed to connect a sequence of numbers as quickly as possible, with total time recorded. Shorter completion times reflect better cognitive performance.
Montreal Cognitive Assessment (MoCA) | Before and inmediately after the intervention
  The MoCA is a comprehensive screening tool for mild cognitive impairment, evaluating domains such as executive function, memory, attention, visuospatial ability, and orientation. The score ranges from 0 to 30. Higher scores reflect better overall cognitive function.
Physical Resilience Instrument for Older Adults (PRIFOR) | Before and inmediately after the intervention
  The Physical Resilience Instrument for Older Adults (PRIFOR) is a validated 16-item questionnaire designed to assess an individual's capacity to recover and adapt following physical stressors such as illness, injury, or functional decline. It evaluates both internal and external resilience factors across four domains: physical strength and energy, emotional and mental coping ability, perceived control and adaptability, and support from social and healthcare systems. Each item is rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree), producing a total score ranging from 16 to 80. Higher scores reflect greater physical resilience, indicating a stronger ability to maintain or regain function in the face of health challenges.
Timed Up and Go with Manual Task (TUG-M) | Before and inmediately after the intervention
  The TUG-M is a dual-task version of the standard TUG in which participants are asked to perform the same sequence while carrying a cup of water with one hand. This variant assesses functional mobility under motor interference and challenges postural control and attention. Time to complete the task is recorded in seconds. Lower times reflect better motor coordination and dual-task performance, indicating greater safety during daily life activities.
Timed Up and Go with Cognitive Task (TUG-C) | Before and inmediately after the intervention
  The TUG-C assesses functional mobility under cognitive load. Participants complete the standard TUG task while simultaneously performing a cognitive task, such as counting backwards or solving a simple mental calculation (e.g., subtracting by threes). This version evaluates the impact of divided attention on mobility and fall risk. Faster times suggest better cognitive-motor integration and executive function.
Cornell Scale for Depression un Dementia (CSDD) | Before and inmediately after the intervention
  The Cornell Scale for Depression in Dementia (CSDD) will be used to assess depressive symptoms in participants with or without cognitive impairment. The scale consists of 19 items covering mood-related signs, behavioral disturbances, physical signs, cyclic functions, and ideational disturbances. Each item is rated from 0 to 2 (0 = absent, 1 = mild or intermittent, 2 = severe), based on interviews with both the patient and an informant. Total scores range from 0 to 38, with higher scores indicating more severe depressive symptoms. Scores above 10 suggest probable major depression, while scores above 18 are highly indicative of a depressive disorder. Lower scores represent better psychological well-being.
Self-reported Vision | Before and inmediately after the intervention
  Self-reported vision will be assessed through a single-item question asking participants to rate their visual ability. Responses are scored as follows: 0 = severe difficulty or complete blindness, 0.5 = mild to moderate difficulty, and 1 = no difficulty. Higher scores indicate better sensory function.
Self-reported Hearing | Before and inmediately after the intervention
  Self-reported hearing will be assessed through a single-item question asking participants to rate their hearing ability. Responses are scored as follows: 0 = severe difficulty or complete deafness, 0.5 = mild to moderate difficulty, and 1 = no difficulty. Higher scores indicate better sensory function.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Francisco Lisón Párraga, Dr, Principal Investigator — Cardenal Herrera University
Locations (1):
- Universidad Ceu Cardenal Herrera, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided